CLINICAL TRIAL: NCT05974904
Title: Association of High-sensitivity C-reactive Protein to Albumin Ratio with Metabolic Dysfunction-associated Fatty Liver Disease and Liver Fibrosis: a Cross-sectional Study
Brief Title: Association of HsCAR with MAFLD and Liver Fibrosis: a Cross-sectional Study
Status: Recruiting | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Tingqiu Wang, Principal Investigator, Chongqing Medical University
Other Study IDs: ChongqingMUU
Record Dates: First submitted 2023-07-21; First posted 2023-08-03 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Metabolic Dysfunction-associated Fatty Liver Disease; Hepatic Steatosis; Liver Fibrosis
Keywords: high-sensitivity C-reactive protein to albumin ratio; metabolic dysfunction-associated fatty liver disease; National Health and Nutrition Examination Survey; control attenuation parameter; liver stiffness measurement; inflammation
MeSH Terms: conditions — Fatty Liver; Liver Cirrhosis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Medical history electronic data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Non-MAFLD group: controlled attenuation parameter<274 dB/m
- MAFLD group: controlled attenuation parameter ≥ 274 dB/m
  Interventions: Other: high-sensitivity C-reactive protein to albumin ratio
- Non-fibrosis group: liver stiffness measurement < 8.2 kPa
- Fibrosis group: liver stiffness measurement ≥ 8.2 kPa
  Interventions: Other: high-sensitivity C-reactive protein to albumin ratio

INTERVENTIONS:
Other: high-sensitivity C-reactive protein to albumin ratio — High-sensitivity C-reactive protein to albumin ratio is an inflammatory indicator which can make a determination of disease severity.
  Groups: Fibrosis group; MAFLD group

SUMMARY:
The goal of this observational study is to investigate the associations between a novel inflammatory marker, high sensitivity C-reactiveprotein to albumin ratio (hsCAR), and steatosis and fibrosis of metabolic dysfunction-associated fatty liver disease (MAFLD).

The main question[s] it aims to answer are:

[question 1] Can hsCAR serve as a clinical indicator to determine whether a patient has MAFD? [question 2] Can hsCAR determine whether MAFLD patients are complicated with liver fibrosis?

DETAILED DESCRIPTION:
Background Inflammation is related to the occurrence and development of fatty liver. Our research aimed to investigate the link between an inflammatory indicator, high-sensitivity C-reactive protein to albumin ratio (hsCAR), and metabolic dysfunction-associated fatty liver disease (MAFLD).

Methods Ultrasonic indices were used to evaluate the severity of liver steatosis and fibrosis of participants from the NHANES database, respectively. The relationship between hsCAR and MAFLD was explored using multivariate logistic regression analysis, restricted cubic splines (RCS) as well as threshold analysis. Finally, subgroup analyses were performed using the same methodology.

ELIGIBILITY:
Inclusion Criteria:

* Total participants from NHANES 2017-2020
* Participants diagnosed with MAFLD. Metabolic dysfunction-associated fatty liver disease (MAFLD) is the term used to describe hepatic steatosis in the presence of metabolic abnormalities, excess weight, obesity, or type 2 diabetic mellitus.

  1. Diagnosis of diabetes mellitus: (1) taking glucose-lowering drugs; (2) HbA1c ≥ 6.5% (48 mmol/mol); (3) fasting plasma glucose ≥ 7.0 mmol/L (126 mg/dL); (4) 2-hour plasma glucose (2hPG) ≥ 11.1 mmol/L (200 mg/dL).
  2. Overweight or obesity: defined as BMI≥25 kg/m2 in Caucasians or BMI≥23 kg/m2 in Asians
  3. If presence of at least two metabolic risk abnormalities:

     * Waist circumference≥102/88 cm in Caucasian men and women (or≥90/80 cm in Asian men and women)
     * Blood pressure≥130/85 mmHg or specific drug treatment
     * Plasma triglycerides≥150 mg/dl (≥1.70 mmol/L) or specific drug treatment
     * Plasma HDL-cholesterol <40 mg/dl (<1.0 mmol/L) for men and <50 mg/dl (<1.3 mmol/L) for women or specific drug treatment
     * Prediabetes (i.e., fasting glucose levels 100 to 125 mg/dl [5.6 to 6.9 mmol/L], or 2-hour post-load glucose levels 140 to 199 mg/dl [7.8 to 11.0 mmol] or HbA1c 5.7% to 6.4% [39 to 47 mmol/mol])
     * Homeostasis model assessment of insulin resistance score≥2.5
     * Plasma high-sensitivity C-reactive protein level >2 mg/L

Exclusion Criteria:

* Liver ultrasound data not available
* participants without complete clinical data
* participants under 18 years old
* participants with cancer.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: They all come from the National Health and Nutrition Examination Survey, which is a database that contains information about demographics, dietary, examination, laboratory and questionnaire of the American population obtained through sophisticated sampling strategies.
Sampling Method: Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
Controlled attenuation parameter | at baseline
  Controlled attenuation parameter is an ultrasound indicator measured by FibroScan to evaluate the degree of liver steatosis

SECONDARY OUTCOMES:
Liver stiffness measurement | at baseline
  Liver stiffness measurement is an ultrasound indicator measured by FibroScan to evaluate the degree of liver stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Tingqiu Wang, Bachelor, Study Director — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eslam M, Newsome PN, Sarin SK, Anstee QM, Targher G, Romero-Gomez M, Zelber-Sagi S, Wai-Sun Wong V, Dufour JF, Schattenberg JM, Kawaguchi T, Arrese M, Valenti L, Shiha G, Tiribelli C, Yki-Jarvinen H, Fan JG, Gronbaek H, Yilmaz Y, Cortez-Pinto H, Oliveira CP, Bedossa P, Adams LA, Zheng MH, Fouad Y, Chan WK, Mendez-Sanchez N, Ahn SH, Castera L, Bugianesi E, Ratziu V, George J. A new definition for metabolic dysfunction-associated fatty liver disease: An international expert consensus statement. J Hepatol. 2020 Jul;73(1):202-209. doi: 10.1016/j.jhep.2020.03.039. Epub 2020 Apr 8. PMID 32278004
- [Background] Eddowes PJ, Sasso M, Allison M, Tsochatzis E, Anstee QM, Sheridan D, Guha IN, Cobbold JF, Deeks JJ, Paradis V, Bedossa P, Newsome PN. Accuracy of FibroScan Controlled Attenuation Parameter and Liver Stiffness Measurement in Assessing Steatosis and Fibrosis in Patients With Nonalcoholic Fatty Liver Disease. Gastroenterology. 2019 May;156(6):1717-1730. doi: 10.1053/j.gastro.2019.01.042. Epub 2019 Jan 25. PMID 30689971
- [Background] Karimi A, Shobeiri P, Kulasinghe A, Rezaei N. Novel Systemic Inflammation Markers to Predict COVID-19 Prognosis. Front Immunol. 2021 Oct 22;12:741061. doi: 10.3389/fimmu.2021.741061. eCollection 2021. PMID 34745112